CLINICAL TRIAL: NCT03189667
Title: Drug Coated Balloons vs Plain Balloons for the Management of Dysfunctional Dialysis Fistula
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment and recent concerns of safety of Paclitaxel coated balloons and associated increased risk death
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC16/035/R
Record Dates: First submitted 2017-06-01; First posted 2017-06-16 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Dysfunctional Dialysis Arteriovenous Fistula
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Intervention Model Description: Open label randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Drug coated balloon angioplasty (Experimental): * Vessel preparation with Pre dilatation
  * Vessel treatment with Drug-coated balloon
  Interventions: Device: Vessel preparation with angioplasty; Device: Drug coated balloon angioplasty
- Plain balloon angioplasty (Active Comparator): * Vessel preparation with Pre dilatation
  * Vessel treatment with additional Plain balloon angioplasty:
  Interventions: Device: Vessel preparation with angioplasty; Device: Plain balloon angioplasty

INTERVENTIONS:
Device: Vessel preparation with angioplasty — Vessel preparation with Pre dilatation:
  * All lesions to be predilated with high pressure balloons until waist is obliterated.
  * At least two minutes dilatation.
  * Balloon sizing: not to exceed the average diameter of adjacent normal appearing non-aneurysmal segments by more than 25%.
  * Multiple lesions:
    * To be treated with single balloon if possible.
    * To be treated with multiple inflation if cannot be covered with single balloon.
Device: Plain balloon angioplasty — Plain balloon angioplasty
  * Vessel treatment with additional Plain balloon angioplasty:
  * Inflation to nominal pressure for at least 1 minute.
  * Balloon size: similar to predilation balloon.
  Arms: Plain balloon angioplasty
Device: Drug coated balloon angioplasty — Lutonix® Drug Coated Balloon: The balloon is coated with a specialized formulation that includes the drug, paclitaxel. The paclitaxel coating is evenly distributed across the working length of the balloon at a surface concentration of 2 μg/mm2. The key functional characteristic of the formulation is to allow for release of paclitaxel to the tissue of the vascular wall during inflation.
  * Inflation to nominal pressure for at least 1 minute.
  * Balloon size: similar to the predilation balloon.
  * New drug coated balloon will be required for each lesion.
  Arms: Drug coated balloon angioplasty

SUMMARY:
Compare the effectiveness of drug-coated balloons to plain balloon angioplasty in reducing stenosis rates in dialysis arteriovenous fistulas (AVFs).

DETAILED DESCRIPTION:
Objectives of the Study:

Hypothesis: Drug-coated balloons improve functional and patency outcomes of failing/dysfunctional hemodialysis fistulas compared to plain uncoated balloons

Aim of the Study:

Compare the effectiveness of drug-coated balloons to plain balloon angioplasty in reducing stenosis rates in dialysis AVFs.

Specific Objectives:

Primary functional endpoint: Access circuit patency based on functional criteria at 12 month.

Primary safety endpoint: Peri procedural complication rate

Secondary endpoints:

* Technical success (<30% residual stenosis without postdilation)
* Access circuit dysfunction free survival (Time to event) based on functional criteria
* Target lesion restenosis free survival (Time to event) (in case of new lesion causes circuit dysfunction)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  * >18 year old
  * Dysfunctional dialysis fistula
* Radiocephalic
* Brachiocephalic
* Brachiobasilic

Clinical criteria for diagnosis of dysfunctional fistula:

* Swelling of the fistula limb
* Prolonged bleeding after withdrawing access needles
* Abnormal pulsations or weak thrill.
* Functional criteria for the diagnosis of dysfunctional criteria:
* Arteriovenous fistula is unable to deliver dialysis blood flow (Qb) of equal to or more than 300 ml/min and/or access recirculation of more than 10% on at least two occasions,
* A rising trend of venous pressure or excessive negative arterial pressure, and/or unable to deliver a Kt/v of 1.2 or more.
* Non-thrombosed

Exclusion Criteria:

* Dysfunctional arteriovenous (AV) grafts
* Thrombosed fistulas
* Intra-stent stenosis
* Stenoses not responding to balloon angioplasty and requiring stenting.
* Stenosis less than 50%
* Surgical intervention that excludes the treatment segment from the access circuit
* Systemic or local (to the fistula) infection treated for less than 10 days prior to the study procedure
* Location of isolated stenosis central to the thoracic inlet.
* Women who are breastfeeding, pregnant or are intending to become pregnant
* Known hypersensitivity or contraindication to contrast medium which cannot be adequately premeditated.
* Sensitivities to heparin, aspirin, other anticoagulant/antiplatelet therapies, and/or paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
AVF circuit patency | 12 month
  Dialysis adequacy to be assessed based on functional criteria

SECONDARY OUTCOMES:
Technical success | intra procedural
  <30% residual stenosis without postdilation
Access circuit dysfunction free survival | 12 month
  Time to event based on functional criteria
Target lesion restenosis free survival | 12 month
  Time to event in case of new lesion causes circuit dysfunction
Number of participants with treatment-related adverse events | 12 month following the procedure
  Number of participants with treatment-related adverse events as assessed by the Society of Interventional Radiology Clinical Practice Guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Arabi, MD, Principal Investigator — King Abdulaziz Medical City
Locations (1):
- King ABdulaziz Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No